CLINICAL TRIAL: NCT03274297
Title: A Randomized, Double-blind, 2-Way Crossover Bioequivalence and Adhesion Study of a Transdermal Contraceptive Patch Manufactured With Newly Sourced Adhesive Components and Currently Marketed EVRA® in Healthy Adult Women
Brief Title: A Study to Evaluate Bioequivalence and Adhesion of a Transdermal Contraceptive Patch Manufactured With Newly Sourced Adhesive Components and Currently Marketed EVRA in Healthy Adult Women
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Janssen Research & Development, LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Other
Other Study IDs: CR108360; 2017-002186-22 (EudraCT Number); RWJ10553CON4001 (Other: Janssen Research & Development, LLC)
Record Dates: First submitted 2017-09-05; First posted 2017-09-06 (Actual); Last update posted 2025-02-03 (Actual); Status verified 2025-01

CONDITIONS: Healthy

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Group 1: Sequence AB (Right/Left) (Experimental): A single patch of currently marketed EVRA patch (Treatment A) will be applied to the right buttock of participants on Day 1 of treatment period 1, followed by application of a single patch of transdermal contraceptive using the newly sourced adhesive component HMW PIB (Treatment B) to left buttock of participants on Day 1 of treatment period 2. The treatment periods will be separated by a washout period of 21 days.
  Interventions: Drug: EVRA patch (NGMN+EE) (Treatment A) (Reference); Drug: HMW PIB patch (NGMN+EE) (Treatment B) (Test)
- Group 2: Sequence BA (Right/Left) (Experimental): Treatment B will be applied to the right buttock of participants on Day 1 in Period 1 followed by Treatment A to the left buttock on Day 1 in Period 2. The treatment periods will be separated by a washout period of 21 days.
  Interventions: Drug: EVRA patch (NGMN+EE) (Treatment A) (Reference); Drug: HMW PIB patch (NGMN+EE) (Treatment B) (Test)
- Group 3: Sequence AB (Left/Right) (Experimental): Treatment A will be applied to the left buttock of participants on Day 1 in Period 1 followed by Treatment B to the right buttock on Day 1 in Period 2. The treatment periods will be separated by a washout period of 21 days.
  Interventions: Drug: EVRA patch (NGMN+EE) (Treatment A) (Reference); Drug: HMW PIB patch (NGMN+EE) (Treatment B) (Test)
- Group 4: Sequence BA (Left/Right) (Experimental): Treatment B will be applied to the left buttock of participants on Day 1 in Period 1 followed by Treatment A to the right buttock on Day 1 in Period 2. The treatment periods will be separated by a washout period of 21 days.
  Interventions: Drug: EVRA patch (NGMN+EE) (Treatment A) (Reference); Drug: HMW PIB patch (NGMN+EE) (Treatment B) (Test)

INTERVENTIONS:
Drug: EVRA patch (NGMN+EE) (Treatment A) (Reference) — A single transdermal contraceptive patch of EVRA (NGMN + EE) containing 6 milligram (mg) of the progestin NGMN and 600 microgram (mcg) of the EE will be applied to the buttock (right or left) of participants on Day 1 of each treatment period and is removed 7 days after patch application, ie, on Day 8.
  Other Names: RWJ10553
Drug: HMW PIB patch (NGMN+EE) (Treatment B) (Test) — A single transdermal contraceptive HMW PIB (NGMN + EE) patch containing 6 mg of the progestin NGMN and 600 mcg of the EE will be applied to the buttock (right or left) of participants on Day 1 of each treatment period and is removed 7 days after patch application, ie, on Day 8.
  Other Names: RWJ10553

SUMMARY:
The purpose of this study is to determine the bioequivalence of the hormones (ie, norelgestromin [NGMN] and ethinyl estradiol [EE]) from the transdermal contraceptive patch and to evaluate the adhesion of the transdermal contraceptive patch using the newly sourced adhesive component, as compared to the currently marketed EVRA patch.

ELIGIBILITY:
Inclusion Criteria:

* Participant has a body mass index (BMI) between 18 and 30 kilogram per meter square (kg/m^2), inclusive, and body weight not to exceed 100 kilogram
* Participant must be healthy on the basis of physical examination, medical history, vital signs, and 12-lead electrocardiogram (ECG) performed at screening. This will be documented and signed by the investigator in the source document
* Participant must have a negative serum (beta-human chorionic gonadotropin) pregnancy test at screening and negative urine pregnancy tests on Day -1 of each treatment period
* Participant must be willing and able to adhere to the prohibitions and restrictions specified in this protocol
* Participant must be surgically sterile with intact ovaries, abstinent, or, if sexually active, be practicing an effective method of non-hormonal birth control (example [eg], intrauterine device [IUD], double barrier method, male partner sterilization) before admission and throughout the study

Exclusion Criteria:

* Participant has a history of or current clinically significant medical illness including (but not limited to) cardiac arrhythmias or other cardiac disease, hematologic disease, coagulation disorders (including any abnormal bleeding or blood dyscrasias), lipid abnormalities, significant pulmonary disease, including bronchospastic respiratory disease, diabetes mellitus, renal or hepatic insufficiency, thyroid disease, neurologic or psychiatric disease, infection, cholelithiasis (gall stone disease), chronic idiopathic jaundice, family history of cholestatic jaundice, or any other illness that the investigator considers should exclude the participant or that could interfere with the interpretation of the study results
* Participant has clinically significant abnormal values for hematology, biochemistry, or urinalysis at screening as deemed appropriate by the investigator
* Participant has abnormal thyroid stimulating hormone level at screening
* Participant has clinically significant abnormal 12-lead ECG, vital signs, or physical examination at screening as deemed appropriate by the investigator
* Participant has a history or presence of disorders commonly accepted as contraindications to sex hormonal therapy including, but not limited to, the following: a) Deep vein thrombophlebitis or thromboembolic disorders; b) Cerebral vascular or coronary artery disease, chronic untreated hypertension, or migraines; c) Benign or malignant liver tumor that developed during the use of oral contraceptives or other estrogen-containing products; d) Known or suspected estrogen-dependent neoplasia

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 70 (Actual)
Dates: Start 2017-09-20 (Actual); Primary Completion 2018-05-07 (Actual); Study Completion 2018-05-07 (Actual)

PRIMARY OUTCOMES:
Mean Steady-State Concentration (Css) for Norelgestromin (NGMN) | 48 to 168 hours post-dose
  Mean steady-state concentration for NGMN after patch application, will be calculated as the mean concentration between 48 hours and 168 hours after patch application.
Mean Steady-State Concentration (Css) for Ethinyl Estradiol (EE) | 48 to 168 hours post-dose
  Mean steady-state concentration for EE after patch application, will be calculated as the mean concentration between 48 hours and 168 hours after patch application.
Area Under the Plasma Concentration-Time Curve From Time 0 (Patch Application) to Time 168 hours Post-dose (AUC[0-168]) for NGMN | Pre-dose to 168 hours post-dose
  Area under the concentration versus time curve from zero (patch application) to 168 hours of NGMN in plasma will be assessed.
Area Under the Plasma Concentration-Time Curve From Time 0 (Patch Application) to Time 168 hours Post-dose (AUC[0-168]) for EE | Pre-dose to 168 hours post-dose
  Area under the concentration versus time curve from zero (patch application) to 168 hours of EE in plasma will be assessed.
Area Under the Plasma Concentration-Time Curve From Time 0 (Patch Application) to Time 240 hours Post-dose (AUC[0-240]) for NGMN | Pre-dose to 240 hours post-dose
  Area under the concentration versus time curve from zero (patch application) to 240 hours of NGMN in plasma will be assessed.
Area Under the Plasma Concentration-Time Curve From Time 0 (Patch Application) to Time 240 hours Post-dose (AUC[0-240]) for EE | Pre-dose to 240 hours post-dose
  Area under the concentration versus time curve from zero (patch application) to 240 hours of EE in plasma will be assessed.
Area Under the Plasma Concentration-Time Curve From Time 0 (Patch Application) to Infinite Time (AUC[0-infinity]) for NGMN | Pre-dose to 240 hours post-dose
  Area under the concentration versus time curve from zero (patch application) to infinite time of NGMN in plasma will be assessed.
Area Under the Plasma Concentration-Time Curve From Time 0 (Patch Application) to Infinite Time (AUC[0-infinity]) for EE | Pre-dose to 240 hours post-dose
  Area under the concentration versus time curve from zero (patch application) to infinite time of EE in plasma will be assessed.
Cumulative Adhesion Percentage Ratio | Baseline (Day 1) and every 24 hours after patch application up to patch removal at 168 hours (Day 8)
  Adhesion of patches will be assessed in accordance with the European Medicines Agency (EMA) 0-5 scoring system. An estimated percentage of adhesion, to a whole integer, will be obtained (EMA 0-5 [percentage (%)] scoring). Estimated percentages of adhesion and corresponding EMA 0-5 score at each interval will be recorded in each participant's electronic case report form. The scoring system for adhesion of transdermal patches is indicated as follows: 0= greater than (>) 90-100% of the patch area adheres; 1= >80-90% of the patch area adheres; 2= >70-80% of the patch area adheres; 3= >60-70% of the patch area adheres; 4= >50-60% of the patch area adheres; 5= 0-less than or equal to (<=) 50% of the patch area adheres.

SECONDARY OUTCOMES:
Irritation Potential | Screening, pre-dose, 168.5 and 192 hours post-dose
  Percentage of participants with specific application site reactions will be summarized for each treatment.

CONTACTS AND LOCATIONS:
Overall Officials: Janssen Research & Development, LLC Clinical Trial, Study Director — Janssen Research & Development, LLC
Locations (1):
- Clinical Pharmacology Unit, Merksem, Belgium

REFERENCES:
- See also: A Randomized, Double-blind, 2-Way Crossover, Bioequivalence and Adhesion Study of a Transdermal Contraceptive Patch Manufactured With Newly Sourced Adhesive Components and Currently Marketed EVRA® in Healthy Adult Women — https://filehosting-v2.pharmacm.com/api/Attachment/Download?tenantId=80217051&parentIdentifier=CR108360&attachmentIdentifier=d571bf10-3740-4505-8684-14039f9d6a41&fileName=CR108360_CSR.pdf&versionIdentifier=